CLINICAL TRIAL: NCT02891759
Title: A Single-Blinded Randomized Prospective Trial to Compare Outcomes Between Two Acellular Dermal Matrices Used for Immediate, Post-Mastectomy Breast Reconstruction
Brief Title: Compare Outcomes Between Two Acellular Dermal Matrices
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: RTI Surgical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201608168
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Subcutaneous; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Alloderm RTU (Experimental): * Prior to the date of mastectomy, the BREAST Q patient-reported outcome survey will be administered for routine clinical care purposes. It may occur before or after enrollment.
  * On the day of surgery, patients will receive standardized preoperative care, a skin- or nipple-sparing mastectomy from an experienced surgical breast oncologists and immediate tissue expander breast reconstruction with Dr. Myckatyn or Dr. Tenenbaum. Uniform operative techniques will be used in both treatment groups. All patients will receive either a 16x8 cm (128 sq cm) ADM graft for postpectoral reconstruction or 16x20 cm (320 sq cm) for prepectoral reconstruction. Patients randomized to Group A will receive Alloderm RTU
  * A post-operative version of the Breast Q validated in patients who have received tissue expanders will be administered between 1 and 3 months after tissue expander insertion, and again prior to exchange for an implant or flap (or at time of patient-requested removal
  Interventions: Other: Alloderm RTU; Procedure: Skin or nipple-sparing mastectomy; Other: Breast Q; Procedure: Surgery
- Group B: Cortiva 1mm Allograft Dermis (Experimental): * Prior to the date of mastectomy, the BREAST Q patient-reported outcome survey will be administered for routine clinical care purposes. It may occur before or after enrollment.
  * On the day of surgery, patients will receive standardized preoperative care, a skin- or nipple-sparing mastectomy from an experienced surgical breast oncologists and immediate tissue expander breast reconstruction with Dr. Myckatyn or Dr. Tenenbaum. Uniform operative techniques will be used in both treatment groups. All patients will receive either a 16x8 cm (128 sq cm) ADM graft for postpectoral reconstruction or 16x20 cm (320 sq cm) for prepectoral reconstruction. Patients randomized to Group B will receive Cortiva 1mm Allograft Dermis
  * A post-operative version of the Breast Q validated in patients who have received tissue expanders will be administered between 1 and 3 months after tissue expander insertion, and again prior to exchange for an implant or flap (or at time of patient-requested removal
  Interventions: Other: Cortiva 1mm Allograft Dermis; Procedure: Skin or nipple-sparing mastectomy; Other: Breast Q; Procedure: Surgery

INTERVENTIONS:
Other: Alloderm RTU — -Most commonly used acellular dermal matrices
  Arms: Group A: Alloderm RTU
Other: Cortiva 1mm Allograft Dermis — -Tutoplast processed dermis
  Arms: Group B: Cortiva 1mm Allograft Dermis
Procedure: Skin or nipple-sparing mastectomy — -Standard of care
Other: Breast Q — * 15 questions
  * 10 questions in Part A asking how has the patient been feeling in past 24 hours, answers range from 0-10 with 0=none of the time and 10=all of the time
  * Part B has 5 questions asking patient if she has had any of the following in the last 24 hours, answers ranging from 0-10 with 0=none of the time and 10=all of the time
Procedure: Surgery — * To address the tissue expander
  * Standard of care

SUMMARY:
This study will evaluate the performance of Alloderm RTU medium (LifeCell) vs. Cortiva 1mm Allograft Dermis (RTI Surgical®, Inc.). These are the thinnest versions of acellular dermal matrices (ADM) offered by both vendors and can be used for post-mastectomy breast reconstruction. Alloderm RTU medium has a thickness of 1.6±0.4 mm, while Cortiva 1mm Allograft Dermis has a thickness of 1.0±0.2 mm. In the context of breast reconstruction, these ADMs are used in the same manner. They may be inserted with a tissue expander immediately after skin- or nipple-sparing mastectomy. The investigators will examine breast-reconstruction associated complication rates, pre- and post-operative patient reported outcomes using the Breast Q, and physician reimbursement as well as direct hospital costs. The endpoint will be either exchange of the tissue expander for a permanent breast implant or autologous flap, explantation due to patient preference, development of a complication, or less common reasons. The investigators propose that Cortiva 1mm Allograft Dermis and Alloderm RTU will have equivalent complication and patient reported outcome rates as well as physician reimbursement, but that direct hospital cost will be less with Cortiva 1mm Allograft Dermis.

ELIGIBILITY:
Inclusion Criteria:

* Sex: Females
* Age: 22 to 70 years old
* Preoperative surgical plan: Immediate placement subpectoral (subpectoral and postpectoral are synonymous) tissue expander with ADM or Immediate placement prepectoral tissue expander or implant with ADM
* Mastectomy type: Skin-sparing or nipple-sparing mastectomy with or without sentinel lymph node biopsy; may be unilateral or bilateral mastectomy
* Able to understand and willing to sign IRB approved written informed consent document.

Exclusion Criteria:

-Pregnant and/or breastfeeding.

Ages: 22 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Incidence of premature tissue expander (TE) removal | Up to 15 months
  * All participants meeting the eligibility criteria who have signed a consent form and have a skin- or nipple-sparing mastectomy and immediate tissue expander breast reconstruction will be included in the analyses of the primary study endpoint.
  * A breast with the TE removed before planned exchange to a permanent breast implant is considered to have had a premature TE removal

SECONDARY OUTCOMES:
Patient satisfaction as measured by Breast Q | Up to 15 months
  * Each domain contains separate modules that investigate physical, psychosocial, and sexual well-being as well as their satisfaction with their care, breasts, and overall outcome.
  * It also investigates patient expectations in the preoperative questionnaire, and degree to which expectations were met in the post-operative version.
  * Each module generates a Q-score on a 0-100 scale that can be used for quantitative analysis to enable statistical comparison of the pre- to the post-operative state.
Health related quality of life as measured by Breast Q | Up to 15 months
  * Each domain contains separate modules that investigate physical, psychosocial, and sexual well-being as well as their satisfaction with their care, breasts, and overall outcome.
  * It also investigates patient expectations in the preoperative questionnaire, and degree to which expectations were met in the post-operative version.
  * Each module generates a Q-score on a 0-100 scale that can be used for quantitative analysis to enable statistical comparison of the pre- to the post-operative state.
Duration of drain use | Up to 15 months
  -The number of days a drain is used after surgery
Incidence of analgesic use for pain | Up to 15 months
  -Outpatient analgesia beyond preoperative analgesic requirements will be recorded, and will include no pain medicine, celecoxib, gabapentin, acetaminophen, hydrocodone, oxycodone, OxyContin, ibuprofen, hydromorphone, cyclobenzaprine, and methadone.
Incidence of infection as measured by presence or absence of cellulitis | Up to 15 months
  -The number of participants who experience cellulitis
Incidence of non-infectious complications | Up to 15 months
  -These will include seroma (and method(s) of seroma diagnosis), incisional dehiscence, necrosis of the mastectomy skin flap, dehiscence of the ADM from the chest wall or pectoralis muscle, hematoma, or a pathologic (grade III or IV) capsular contracture.
Nature of second surgery as measured by type of surgery enrolled patients undergo to address their tissue expander after its initial insertion | Up to 15 months
  -Document type of second surgery each participants has after their initial tissue expander
Degree of acellular dermal matrices (ADM) incorporation | Up to 15 months
  -A qualitative scale, from 1-4 will be used to quantity ADM incorporation. This will be recorded upon inspection of the ADM at the time that the tissue expander is readdressed.
Comparison of direct hospital costs | Up to 15 months
  -These are available through Barnes hospital and will be normalized to Medicare rates by conversion from relative value units (RVU) due to heterogeneity in payer mix. Line item costs as well as patient-level data will not be available due to the proprietary nature of these products. However, normalized, aggregate patient data for the cycle of care in each study arm (Alloderm RTU vs Cortiva 1mm Allograft Dermis) is available and will be calculated. "Direct costs" are those that can be traced directly to a department, product or service, excluding overhead costs, and thus reflect the hospital's assessment of the cost it incurred providing the specific services and supplies used by the patients. All breast reconstruction related costs performed by Barnes, or Barnes West County hospital from the first surgery up until immediately before the second surgery will be included.
Comparison of physician reimbursements | Up to 15 months
  -These are available through the Department of Surgery and will be normalized to Medicare rates by conversion from relative value units (RVU) due to heterogeneity in payer mix. Line item costs as well as patient-level data will not be available due to the proprietary nature of these products. However, normalized, aggregate patient data for the cycle of care in each study arm (Alloderm vs Cortiva 1mm Allograft Dermis) is available and will be calculated. All breast reconstruction related costs billed by Washington University Physicians from the first surgery up until immediately before the second surgery will be included.
Amount of tissue expander fill | At the time of surgery
  -This is breast-level data since the left and right side may differ in bilateral reconstruction cases. The investigators already track tissue expander fills as part of the electronic medical record. The amount of tissue expander fill during surgery and device type are recorded in the operative record.
Immediate implant type as measured by volume (cc) | At the time of surgery
Immediate implant type as measured by manufacturer | At the time of surgery
Immediate implant type as measured by shape | At the time of surgery
Immediate implant type as measured by fill | At the time of surgery
Immediate implant type as measured by surface characteristics | At the time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Terence M Myckatyn, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu